CLINICAL TRIAL: NCT01091623
Title: Effects of Strength Training in Combination With Endurance Training on Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 001/2005
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2005-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: improvement of exercise capacity in patients with COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (3):
- strength training (Active Comparator)
  Interventions: Other: training
- endurance training (Active Comparator)
  Interventions: Other: training
- combined training (Active Comparator)
  Interventions: Other: training

INTERVENTIONS:
Other: training
  Arms: strength training
Other: training
  Arms: endurance training
Other: training
  Arms: combined training

SUMMARY:
Background. Exercise intolerance is one of the most devastating consequences of chronic obstructive pulmonary disease (COPD). Abnormalities in peripheral muscle function such as weakness and reduction in oxidative enzyme activities are commonly found in these patients and may contribute to exercise intolerance.To evaluate whether a systemic weightlifting exercise may improve exercise capacity better than endurance training, or a combined training is more effective, the investigators compared three different training regimens, endurance training alone, systemic weightlifting training alone or a combination of both endurance and weightlifting training.

Methods.36 patients with stable COPD will be evaluated before and after a 4 month training program. Each evaluation include a stepwise exercise test on an ergocycle up to the individual maximal capacity during which minute ventilation (VE), oxygen consumption (VO2), carbon dioxide production (VCO2), and arterial lactic acid concentration will be measured and the peripheral muscle strength will be determined with the one repetition maximum for eight different muscle groups. Percutaneous needle muscle biopsy from the M.vastus lateralis will be performed before and after the training period in order to determine the fiber-type proportions. Patients are assigned to one of the following three groups (1) endurance training consisted of 20 min exercise sessions on a calibrated ergocycle two times a week, with a target training intensity at 60% of individual maximum oxygen uptake, (2) systemic weightlifting training two times a week with eight different exercises, each session consist of 15 repetitions of each muscle group, (3) combination of endurance training and systemic weightlifting training.

Statistical analysis. Baseline data for all patients enrolled in the study will be compared by one-way analysis of variance for the three study groups. Results before and after training will be analyzed by two- way analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

1. age: 40-75 years
2. mild to moderate COPD patients according to the staging schemata of the austrian society of lung and tuberculosis disease (ÖGLUT)

Exclusion Criteria:

1. acute infection
2. reduced left ventricular function
3. myocardial infarction
4. stroke
5. severe pulmonary hypertension (mpap>40mmHg)
6. insufficient treated hypertension RR>160/95) (participation with sufficient treatment )
7. severe cardiac arrhythmia
8. malignant diseases
9. severe osteoporosis
10. nicotine abuses
11. other severe chronic diseases

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
increase of exercise capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Vonbank K, Strasser B, Mondrzyk J, Marzluf BA, Richter B, Losch S, Nell H, Petkov V, Haber P. Strength training increases maximum working capacity in patients with COPD--randomized clinical trial comparing three training modalities. Respir Med. 2012 Apr;106(4):557-63. doi: 10.1016/j.rmed.2011.11.005. Epub 2011 Nov 26. PMID 22119456